CLINICAL TRIAL: NCT04159610
Title: A Randomized, Open-Label, Multiple Dose, Two-Period Crossover Study Evaluating Maximum Use 1% GPB Cream Versus Qbrexza® (Glycopyrronium) Cloth 2.4% in Men and Women with Primary Axillary Hyperhidrosis
Brief Title: Assessment of Safety, Tolerability and Efficacy of 1% GPB Cream Versus Qbrexza® (Glycopyrronium) Cloth 2.4% Under Maximum-Use Conditions in Subjects with Primary Axillary Hyperhidrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was not pursued for internal reasons
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GPBBr-02/2019
Record Dates: First submitted 2019-09-09; First posted 2019-11-12 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2021-08

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Excessive sweating
MeSH Terms: conditions — Hyperhidrosis | interventions — glycopyrronium tosylate; Glycopyrrolate; Textiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- WO 3970 (Experimental): Formulation containing WO 3970 for topical application
  Interventions: Drug: WO3970
- Qbrexza® (glycopyrronium) cloth, 2.4%, for topical use (Active Comparator): Qbrexza® (glycopyrronium) cloth, 2.4%, for topical use
  Interventions: Drug: Qbrexza® (glycopyrronium) cloth, 2.4%, for topical use

INTERVENTIONS:
Drug: WO3970 — Application of cream to each axilla
  Arms: WO 3970
Drug: Qbrexza® (glycopyrronium) cloth, 2.4%, for topical use — Qbrexza should be applied to the clean, dry, intact skin, of your underarm areas only
  Arms: Qbrexza® (glycopyrronium) cloth, 2.4%, for topical use

SUMMARY:
The aim of this study is to investigate the safety, tolerability and efficacy of 1% GPB Cream compared to Qbrexza® (glycopyrronium) cloth, 2.4%, for topical use under maximum use conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe primary axillary hyperhidrosis with a HDSS score of 3 or 4
* At least 50 mg of sweat production in each axilla measured gravimetrically at room temperature and at a humidity consistent with the normal climate in that area over a period of 5 minutes (patients should have acclimatized to that room for at least 30 minutes)
* Men and women aged 18 to 65 years at the time of informed consent with a body mass index of 18-32 kg/m2
* Able to comply with protocol requirements, including overnight stays, blood sample collections as defined in the protocol subjects
* Willing and able to provide written informed consent

Exclusion Criteria:

* Known allergy to any of the components in the investigational product.
* Hypersensitivity against glycopyrrolate
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria, climacteric hyperhidrosis.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Botulinum toxin treatment in the prior 4 months.
* Angle closure glaucoma or its precipitation (narrow angle).
* Mycotic, other skin infections and other dermal disorder including infection at anticipated application sites in either axilla.
* Any condition or situation that, in the investigator's or sub-investigator's opinion, may interfere with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Steady State systemic Levels of glycopyrronium | Day-1, Day 1 to Day 13, Day 16

SECONDARY OUTCOMES:
Systemic pharmacokinetic profile of glycopyrronium at steady state (Area under the drug concentration time curve (AUC)) | Day -1, Day 1 to 13, Day 16
Systemic pharmacokinetic profile of glycopyrronium at steady state (Maximum concentration (Cmax)) | Day -1, Day 1 to 13, Day 16
Systemic pharmacokinetic profile of glycopyrronium at steady state (Time to CMax (Tmax)) | Day -1, Day 1 to 13, Day 16
Systemic pharmacokinetic profile of glycopyrronium at steady state (Elimination half-life (t1/2)) | Day -1, Day 1 to 13, Day 16
Adverse events (AEs) | Day -1 of study period 1 to Day 16
Clinical chemistry | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  Albumin, alkaline phosphatase, ALT, AST, BUN, calcium, chloride, CO2, creatinine, direct bilirubin, GGT, glucose, LDH (lactate dehydrogenase), phosphorus, potassium, sodium, total bilirubin, total cholesterol, total protein, uric acid
Hematology | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  Hematocrit, hemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, differentials (neutrophils, eosinophils, basophils, lymphocytes, and monocytes), platelet count, and reticulocytes
Urinalysis | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  Color, specific gravity, pH, glucose, ketones, protein, bilirubin, urobilinogen, WBCs, RBCs, and microscopy
BP | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  mmHg
Respiratory rate | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  breaths per minute
Temperature | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  °C
Heart rate | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  bpm
12-lead ECG | Screening, Day 1-13 of study period 1 and period 2
  beats per minute [bpm], PR, QRS, QT, QTc, QTcF, and QTcB interval
Physical examination | Screening, Day -1, Day 16
  General appearance; eyes; ears, nose and throat; head and neck; chest and lungs; cardiovascular; Abdomen; musculoskeletal; lymphatic; dermatological; neurological and extremities
Local tolerability | Day -1, Day 1-13, Day 16 of study period 1 and period 2
  Dermal Evaluation of erythema, edema and papules
Sweat production by gravimetric measurement | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  5-minute measurement [filter paper] interval first without then repeated with an immediately preceded subject consumption of 250 mL of hot water swallowed within 1 minute
Hyperhidrosis Disease Severity Scale (HDSS) | Screening, Day -1, Day 1 to 13, Day 16 of study period 1 and period 2
  The Hyperhidrosis Disease Severity Scale (HDSS) is a disease-specific, quick, and easily-understood diagnostic tool that provides a qualitative measure of the severity of the patient's condition based on how it affects daily activities. HDSS is a four item scale. A score of 1 or 2 indicates mild or moderate Hyperhidrosis. A score of 3 or 4 indicates severe Hyperhidrosis.
Hyperhidrosis Quality of Life Questionnaire (HydroQoL) | Day -1, Day 1 to 13 of period 1 and period 2
  Hyperhidrosis Quality of Life Questionnaire (HydroQoL) is an 18-item, validated, Patient reported Outcome Hyperhidrosis Quality of life Instrument. It is devided into 2 Domains: A Daily Life Activities Domain (6 items) and a Psychosocial Domain (12 items). The items are scored on a 3-point scale (0=no, not at all, 1=a Little, 2=very much).